CLINICAL TRIAL: NCT05576831
Title: STRatIfication of Vulvar Squamous Cell Carcinoma by HPV and p53 Status to Guide Excision: STRIVE Study
Brief Title: STRatIfication of Vulvar Squamous Cell Carcinoma by HPV and p53 Status to Guide Excision
Acronym: STRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Gynecologic Cancer Initiative (Other); Australia New Zealand Gynaecological Oncology Group (Other); Canadian Cancer Trials Group (Network)
Responsible Party: Principal Investigator, Jessica McAlpine, Co-Division Head, Gynecologic Oncology Professor, Department of Obstetrics and Gynecology Gynecologic Tissue Bank Director, British Columbia Cancer Agency
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRIVE
Record Dates: First submitted 2022-10-01; First posted 2022-10-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Vulvar Cancer
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV-A VSCC (No Intervention): Patients with HPV-A VSCC and margins that are negative for cancer but <8mm (regardless of in-situ (HSIL) margin status) will be eligible for the de-escalation prospective study.
- HPV-I VSCC (Experimental): If the margins are negative for cancer but <8mm, or positive for Differentiated vulvar intraepithelial neoplasia (dVIN), and/or positive for p53 abnormality on IHC, these patients will be randomized (2:1) to further re-excision vs observation only.
  Interventions: Procedure: Re-excision

INTERVENTIONS:
Procedure: Re-excision — Re-excise (one take back only) Excise scar aiming for 1-2cm margin
  Arms: HPV-I VSCC

SUMMARY:
Vulvar cancer affects the external genitalia of women. This type of cancer is uncommon, arising mostly in older women and has been neglected in research and clinical trials. Over the recent years, investigators have learned that the most common type of vulvar cancer; vulvar squamous cell carcinoma (VSCC) develops from pre-cancerous lesions via different pathways. One pathway is associated with human papillomavirus (HPV) infection, and another is related to chronic inflammatory skin conditions (and not HPV). The VSCCs arising from these two principal pathways; HPV- associated (HPV A) and HPV-independent (HPV I), behave differently with different risks of recurrence, and different response to treatments. HPV-I VSCC are further defined by mutations in TP53 (Tumor Protein 53), which identify a group of patients with aggressive disease. Currently treatment is the same for all women with vulvar cancer, and consequently many women may be overtreated, and many women are not treated enough. Given evolving knowledge of this disease, this 'one size fits all' approach may no longer be appropriate. The investigators aim in this study is to see if personalizing surgical therapy for patients with vulvar cancer based on HPV and TP53 status will improve outcomes.

DETAILED DESCRIPTION:
Purpose:

The aim of this prospective study is to determine if implementation of HPV(p16) and p53 stratified management algorithms will improve outcomes for women with VSCC.

Hypothesis:

Primary:

Molecular stratification of VSCC, using margin status for both HPV and p53 pathology to direct surgical management, will improve clinical outcomes.

Patient Reported Outcomes (PRO) Hypothesis:

In women with HPV-associated (HPV-A) VSCC who undergo less radical surgery, treatment-related side effects will be reduced, health-related quality of life will be improved, and fear of cancer recurrence will not be increased, when compared to patients who undergoing standard surgery. PROs that are expected to be improved in this subgroup are: satisfaction with body image, frequency and enjoyment of sexual activity, urinary symptoms, and genital pain. In women with HPV-independent (HPV-I) VSCC, the expected PRO/HRQL (Health-related quality of life) trajectory is expected to remain unchanged in the intervention group compared to the observation group, and fear of recurrence will be decreased.

Justification:

Most VSCC guidelines today recommend tumour-free pathological margins of 8mm or more to adequately treat the primary tumour. These guidelines are based on retrospective data which did not stratify patients based on HPV or TP53 mutation status.

HPV-I VSCC: there is now data suggesting investigators are undertreating these patients and that surgical margins defined by proximity of invasive disease, presence of preinvasive disease and p53 IHC (Immunohistochemistry) status will guide the need for re-excision and optimize local disease control.

Goal in HPV-I VSCC = demonstrating re-excision to achieve clear margins will improve outcomes.

HPV-A VSCC: there is data supporting that investigators are likely overtreating these patients, and the absence of invasive disease at the resection margin will be sufficient without loss of local control and will improve patient reported outcomes.

Goal in HPV-A VSCC= demonstrating de-escalation of surgery is safe(and will improve QoL).

Objectives:

Primary Objective:

To determine if implementation of HPV and p53 stratified algorithms to guide surgical management will improve outcomes in patients with VSCC; based on 3-year local recurrence rates in both HPV-I and HPV-A disease

Secondary Objectives:

1. Determine the health economic impact (EQ-5D) of implementation of HPV and p53 stratified treatment algorithms
2. Determine the patient reported outcomes (EORTC QLQ (Quality of Life Questionnaire) -C30 and EORTC QLQ-VU34), patient decisional conflict, patient satisfaction /acceptance with HPV and p53 stratified care in VSCC
3. Determine the disease specific survival (DSS) and overall survival (OS) for HPV-I and HPV-A VSCC managed per algorithms
4. Determine the feasibility of implementation of routine p16 and p53 IHC reporting in VSCC pathology (proportion of patients who had p53 and p16 IHC successfully performed in an acceptable turnaround time ie >85% of patients within 21 days of surgery)

RESEARCH DESIGN:

The HPV-I arm of the study will be conducted as a phase II, randomised control trial and the HPV-A arm of the study will be a prospective trial.

STATISTICAL ANALYSIS:

The Kaplan-Meier method will be used to estimate 3-year rates of recurrence-free survival, vulvar cancer-specific survival, and overall survival and associated 95% confidence interval with the events defined as any recurrence or death for recurrence-free survival, death due to vulvar cancer for vulvar cancer-specific survival, and death due to any cause for overall survival. Women without the event observed at the time of analysis will be censored at the last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary diagnosis of vulvar squamous cell carcinoma
* Surgically staged FIGO (International Federation of Gynaecology and Obstetrics) I-II disease
* Margin status after primary surgery:

  * HPV-I VSCC: margins are negative for cancer but <8mm, and/or positive for dVIN, and/or positive for p53 abnormality on IHC
  * HPV-A VSCC: margins are negative for cancer but <8mm (regardless of in-situ (HSIL) margin status)
* Age ≥18 years old
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate. A similar process must be followed for sites outside of Canada as per their respective cooperative group's procedures.

Exclusion Criteria:

* Recurrent vulvar squamous cell carcinoma
* Non-squamous cell carcinoma histotypes
* FIGO stage III- IV disease
* Patients referred for adjuvant radiation for close margins
* Margins positive for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2031-11-25 (Estimated); Study Completion 2031-11-25 (Estimated)

PRIMARY OUTCOMES:
Local Vulvar Disease Recurrence - Local vulvar disease recurrence rate (within 3 years) in HPV-I and HPV-A vulvar squamous cell carcinoma | 3 years from study enrollment
  Duration of time from registration to time of recurrent disease in the vulvar

SECONDARY OUTCOMES:
Health Economic Impact of implementation of HPV and p53 stratified treatment algorithms - Measure the delta in surgical parameters (surgical take backs, longer hospital stay for more extensive surgery) | through study completion, an average of 1 year
  Health utility scores will be obtained through multi-attribute quality of life instruments such as the EQ-5D-5L. Outcome measure will be the incremental cost-effectiveness ratio, which is defined as the difference in cost divided by the difference in effectiveness between the 2 treatment strategies.
Patient Reported Outcome EORTC QLQ-C30 - Measures subject's physical, psychological and social functions. | Preoperatively, after surgery at 4-6 weeks, 4 months, 8 months and 12 months, through study completion, an average of 1 year
  Assess the quality of life of cancer patients
Patient Reported Outcome EORTC QLQ-VU34 vulva-specific module - Measures symptoms or problems related to the genital area | through study completion, an average of 1 year
  Assess issues related to the genital area
Patient Decisional Conflict Scale - Change in level of patient decisional conflict is defined as the change in the Decisional Conflict Scale or subscale prior to and after treatment | Preoperative
  a validated tool reflecting patient decision making prior to intervention
Disease-specific survival is defined as the time from study enrolment to the time of death from vulvar cancer. Overall survival is defined as the time from study enrolment to the time of death from any cause. | Every 4 months for first 3 years
  Duration of time from registration to time of death from any cause
Proportion of patients who had p16 IHC and in HPV-I VSCC who had p53 IHC performed on resection margin in an acceptable turnaround time ie >85% of patients tumours had this performed and reported within 21 days of surgery | through study completion, up to 3 years
  proportion of patients who had p53 and p16 IHC successfully performed in an acceptable turnaround time ie >85% of patients within 21 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amy Jamieson, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer - Vancouver Centre, Vancouver, British Columbia, Canada